CLINICAL TRIAL: NCT03298321
Title: Action of the Vidaza on the Atrial Fibrillation
Acronym: AVIFA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0114
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Atrial Fibrillation; Acute Leukemia
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vidaza patients: This study will be performed on adults with Acute Myeloid Leukemia and atrial fibrillation. Only patients treated for the first time with vidaza® within an hospital hematology unit will be included.
  Interventions: Other: Effect of Vidaza treatment

INTERVENTIONS:
Other: Effect of Vidaza treatment — The goal of this study is to evaluate the effects of azacytidine on arrhythmia and left atrium fibrosis.

SUMMARY:
Genomic studies on atrial fibrillation patients have identified polymorphisms in regions surrounding the PITX2 gene, suggesting it could be the locus responsible for atrial fibrillation. The PITX2 gene is essential for establishing the asymmetry between systemic and pulmonary blood flow, which is absolutely required for proper heart functions. In addition, PITX2 is required for the development the atrium myocardium. Investigators have performed transcriptomic analysis on left atrium tissues from atrial fibrillation patients and identify genes whose expression is altered in atrial fibrillation. Among affected genes, PITX2 expression is strongly decreased in the left atrium of atrial fibrillation patients. Moreover, investigators observed that the PITX2 promoter region is hypermethylated in atrial fibrillation patients. Interestingly, DNA methylation is a key actor of gene expression and directly regulates RNA transcription either by directly modulating transcription factor (TF) binding to gene promoters or by modifying local chromatin structures, therefore limiting access of TFs to DNA. These epigenetic modifications are reversible and therefore represent an interesting therapeutic target. Hence, many compounds that inhibit DNA methyl-transferase are currently tested in different disease models. Recently-designed hypomethylating molecules are available, such as the 5'azacytidine (Vidaza®, Celgen Inc.) or the 5-aza-2'-deoxycytidine (Decitabine) (Dacogen®, Janssen Cilag). Investigators have performed preliminary studies on the effect of Decitabine on DNA methylation and proper cardiac function recovering in a SHR model. Results indicate that the chronic delivery of Decitabine improves the arrhythmia profile by reducing tachyarrhythmia, fibrosis, as well as the oxidative stress in SHR left atrium submitted Acute Leukemia is a rare pathology with an incidence of 4 per 100,000 in France. Azacytidine, which is closely related to Decitabine, is commonly used for treating Acute Leukemia and possesses anti-neoplastic effect through multiple mechanisms, including direct cytotoxicity of blood cancer cells and DNA hypomethylation. The goal of this study is to evaluate the effects of azacytidine on arrhythmia and left atrium fibrosis as well, which are the two mains phenotypic manifestation of atrial fibrillation in humans. Investigators hypothesize that azacytidine decreases PITX2 promoter methylation and increases PITX2 expression. Hence, investigators expect to ameliorate the duration of atrium action potential and to observe a decrease of atrium fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient with history of paroxysmal atrial fibrillation, and /or presenting a dilatation of the left atrium.
* Patient selected for a first Vidaza® treatment
* Non-opposition of the patient to participate in the study

Exclusion Criteria:

* Age < 18 years old
* No paroxysmal atrial fibrillation
* Patients with previous history of Vidaza® treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be performed on adults with Acute Myeloid Leukemia and atrial fibrillation. Only patients treated for the first time with vidaza® within an hospital hematology unit will be included.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Evolution of atrial arrhythmic events | Maximum 12 months
  Evolution of the atrial arrhythmic events observed in the inclusion, 6 months or 12 months (according to the frequency of follow-up of the atrial fibrillation) after the beginning of the cure by Holter-ECG.

SECONDARY OUTCOMES:
Evolution of the morphology and the fibrosis atrial | Maximum 12 months
  Evolution of the morphology and the fibrosis atrial observed in the inclusion, 6 months or 12 months (according to the frequency of follow-up of the atrial fibrillation) after the beginning of the cure by transthoracic echocardiography.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service de rythmologie - GH Est-Hôpital Louis Pradel - CHU de Lyon HCL, Bron
  - Centre Léon Berard, Lyon
  - Hopital Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No